CLINICAL TRIAL: NCT06254222
Title: Ethical Crossroads in Nursing Education: Mapping the Terrain of Ethical Sensitivity and Professional Identity Among Nursing Students
Brief Title: Ethical Crossroads in Nursing Education
Status: Active, not recruiting | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Hashem El-Monshed, Associate Professor, Mansoura University
Other Study IDs: ETHICAL12345
Record Dates: First submitted 2024-02-03; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Ethics, Narrative; Professional Identity Formation
MeSH Terms: conditions — Narration; Social Identification

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In conclusion, understanding the variables influencing ethical decision-making among nursing students is crucial for developing interventions to minimize moral distress and promoting their ability to cope with ethical issues and dilemmas. While acknowledging the existence of ethical challenges, it is noteworthy that there is a dearth of studies investigating the intricate relationship between ethical sensitivity and the development of professional identity among nursing students. This research aims to fill this gap, advancing our understanding and providing valuable insights for shaping effective educational practices. In this improvement, the research problem is clearly stated: the need to explore the relationship between ethical sensitivity and professional identity among nursing students, with a call for further research to bridge the existing gap.

In light of the identified research gap regarding the correlation between ethical sensitivity and the development of professional identity among nursing students, this study seeks to answer the following question: How does ethical sensitivity influence the formation of professional identity in nursing students within the context of contemporary healthcare environments, characterized by evolving technology and complex health systems?

ELIGIBILITY:
Inclusion Criteria:

- Participants will be recruited from diverse online communities, including platforms such as Facebook, WhatsApp, and Telegram. The decision to utilize these social media channels is based on their extensive usage within the target population, ensuring effective outreach and active participation. The undergraduate nursing students at the college are expected to establish dedicated social media groups for each academic level.

Exclusion Criteria:

* Students not from nursing background education

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: Nursing students from all levels
Sampling Method: Non-Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-10 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Moral Sensitivity Questionnaire | through study completion, an average of 6 months
  This version was modified by Comrie (2012) to measure the moral sensitivity of student nurses (MMSQSN). According to Comrie, determining the level of ethical sensitivity of student nurses can identify what nursing education programs should do to develop ethical sensitivity. Comrie studied the validity and reliability of the MMSQSN using 250 undergraduate and postgraduate student nurses at a midwestern university. Cronbach's alpha was .64. The MMSQSN is a 7-point Likert type scale that includes 30 items. Statements in the scale are assigned a score between 1 (I completely disagree) and 7 (I completely agree).

SECONDARY OUTCOMES:
Professional Identity Questionnaire | through study completion, an average of 6 months
  This instrument contains 17 items loading on 5 sub-dimensions: professional self-image (6 items), retention benefit and risk of turnover (4 items), social comparison and self-reflection (3 items), career choice independence (2 items) and social modelling (2 items). Items are assessed on a five-point Likert scale ('complete conformity' = 5, 'conformity' = 4, 'neutral' = 3, 'inconformity' = 2, and 'complete inconformity' = 1). The total scores range from 17 to 85, with higher scores indicating a stronger professional identity

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Al Mansurah, Dakhlyia, Egypt

IPD SHARING:
Plan to Share IPD: No